CLINICAL TRIAL: NCT05589220
Title: Multi-method Pilot Study to Evaluate the Interest of Music Therapy Associated to Nicotine Replacement Therapy (NRT) Versus NRT Alone on Craving Related to Smoking Cessation in Students.
Brief Title: Study to Evaluate Music Therapy and Nicotine Replacement Therapy on Craving Related to Smoking Cessation in Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MuSTOPSmok
Record Dates: First submitted 2022-10-04; First posted 2022-10-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
Keywords: prevention; Music Therapy; Craving
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention and NRT (Experimental): The rhythm of the music sessions will be 2 per week in the first month, 1 per week in the second month and 1 every 15 days in the third month. In this group, music intervention will be associated to NRT.
  Interventions: Other: Music Intervention; Drug: Nicotine replacement
- NRT group (Active Comparator): Nicotine Patch, Nicotine Gum As in the intervention group, the physician will adapt the type of NRT according to the patient's smoking profile.
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Other: Music Intervention — Music therapy carried out with MUSIC CARE©
  Arms: Music intervention and NRT
Drug: Nicotine replacement — NRT: Nicotine Patch, Nicotine Gum

SUMMARY:
The study is a randomized, controlled trial comparing music therapy associated to NRT versus NRT alone to evaluate the value of music therapy in improving the management of craving among 120 student smokers (18 to 25 years old). This pilot multi-method study will combine the methodology of clinical trials with qualitative techniques used in social sciences to show the interest of a digital music therapy tool, adapted to a young audience.

DETAILED DESCRIPTION:
The participants will be recruited at the Clinical Investigation Center (CIC) of the University Hospital of Poitiers. At baseline visit, they will be randomly 1:1 assigned to receive either music therapy and NRT or NRT alone for 3 months.

During the 3 months after TQD (Target Quit Date), 3 visits will be performed by practitioners at the CIC. Practitioners will register smoking status of the participant, exhaled carbon monoxide concentration, body weight and all adverse events. Participants will answer questionnaires (FTCQ-12, HAD, MNWS, UPPS).

ELIGIBILITY:
Inclusion Criteria:

* students, age >=18 and <=25 years,
* smoking more than 5 cigarettes per day for at least 6 months,
* motivated to quit smoking,
* without legal tutors or subordination,
* affiliated to a health insurance system as required by the French law on biomedical research,
* written informed consent for participation in the study.

Exclusion Criteria:

* Roommates and couples,
* NRT contraindication
* with depression and/or psychosis and/or cognitive disorder and/or mental retardation,
* substance misuse or alcohol dependence,
* smoking-cessation medication (NRT, bupropion, varenicline) or undergoing cognitive-behavioral therapy or hypnotherapy in the last 3 months,
* electronic cigarette for smoking cessation in the last 3 months,
* Persons benefiting from enhanced protection, i.e. persons deprived of their liberty by a judicial or administrative decision, adults under legal and finally patients in a vital emergency situation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Assess if Music therapy associated to NRT decrease tobacco craving compared to NRT alone | Month 1
  Score of French Version of the Tabacco Craving Questionnaire-12 (FTCQ-12). It consist of 12 questions, each rated on a likert-type scale with 7 response options. Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Test the feasability of such a program in smoking cessation | Month 3
  Music therapy sessions compliance. Number and reasons for not attending music thearpy sessions.
Evaluate the evolution of tobacco craving | Month [2; 3]
  Score of French Version of the Tabacco Craving Questionnaire-12 (FTCQ-12). It consist of 12 questions, each rated on a likert-type scale with 7 response options. Lower scores mean a better outcome.
Evaluate the evolution of Anxiety | Month [1;2; 3]
  HAD (Hospital Anxiety and Depression Scale) score. Maximum score for each score (total A, total D) = 21. Score over 10 definites state of anxiety.
  Lower scores mean a better outcome.
Evaluate the evolution of nicotine withdrawal symptoms | Month [1;2; 3]
  MNWS (Minnesota Nicotine Withdrawal Scale) score. It consist of 8 questions, each rated on a likert-type scale with 0-4 response options. Lower scores mean a better outcome.
Evaluate the evolution of impulsivity | Month [1;2; 3]
  UPPS (Impulsive Behavior Scale) score. It consist of 20 questions, each rated on a likert-type scale with 1-4 response options. Lower scores mean a better outcome.
Evaluate the efficacy of the intervention on smoking cessation | Month [1;2; 3]
  Self reported abstinence or smoking reduction >or=50%

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France